CLINICAL TRIAL: NCT00404131
Title: A Multi-Center, Double-Masked, Randomized, Placebo-Controlled, Dose-Ranging Study of Multiple Ocular Instillations of INS365 Ophthalmic Solution vs. Placebo in Subjects With Dry Eye Disease
Brief Title: Study of INS365 Ophthalmic Solution in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-105
Record Dates: First submitted 2006-11-22; First posted 2006-11-27 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — diquafosol; Ophthalmic Solutions

INTERVENTIONS:
Drug: diquafosol tetrasodium (INS365) Ophthalmic Solution

SUMMARY:
The purpose of this trial is to compare the effectiveness and safety of INS365 Ophthalmic Solution with placebo when applied topically in subjects with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* best corrected visual acuity in both eyes of at least +0.7
* six-month documented history of dry eye disease
* at least mild severity in 2 of the 4 dry eye symptoms
* unanesthetized Schirmer score of less than or equal to 7mm
* corneal fluorescein staining of greater than or equal to 4 (out of 15)

Exclusion Criteria:

* nasally stimulated Schirmer score of less than 3mm in subjects with an initial Schirmer score of 0mm
* ongoing contact lens wear
* current topical ophthalmic medication use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2001-03; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Change in dry eye testing measures and symptoms

SECONDARY OUTCOMES:
Change in dry eye testing measures and symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Amy Schaberg, BSN, Study Director

REFERENCES:
- [Result] Tauber J, Davitt WF, Bokosky JE, Nichols KK, Yerxa BR, Schaberg AE, LaVange LM, Mills-Wilson MC, Kellerman DJ. Double-masked, placebo-controlled safety and efficacy trial of diquafosol tetrasodium (INS365) ophthalmic solution for the treatment of dry eye. Cornea. 2004 Nov;23(8):784-92. doi: 10.1097/01.ico.0000133993.14768.a9. PMID 15502479